CLINICAL TRIAL: NCT00623870
Title: An Open Label Study to Investigate the Maximum Tolerated Dose of RO5045337 in Patients With Acute Myelogenous Leukemia (AML), Acute Lymphocytic Leukemia (ALL), Chronic Myelogenous Leukemia (CML) in Blast Phase, or Refractory Chronic Lymphocytic Leukemia/Small Cell Lymphocytic Lymphoma (CLL / SCLL)
Brief Title: A Study of RO5045337 [RG7112] in Patients With Hematologic Neoplasms.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO21279
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RO5045337

INTERVENTIONS:
Drug: RO5045337 — Multiple ascending doses

SUMMARY:
This study will determine the maximum tolerated dose of RO5045337 and the optimal associated 4 weekly dosing schedule of RO5045337, administered as monotherapy in patients with hematologic neoplasms. A first cohort of patients will receive the starting dose of 20mg/m2/day orally, once daily for 10 days in each 28 day cycle. Subsequent cohorts of patients will receive dose escalations, and possible changes in dosing schedule, based on tolerability and pharmacokinetic knowledge gained from prior treatment cohorts. Different formulations of RO5045337 will be tested and the food effect evaluated. The anticipated time on study treatment is until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >=18 years of age
* Acute myeloid leukemia, acute lymphocytic leukemia, chronic myelogenous leukemia in blast phase, refractory chronic lymphocytic leukemia/small cell lymphocytic lymphoma
* Relapsed or refractory to approved therapies, or no viable alternative therapy available
* ECOG performance status of 0-2

Exclusion Criteria:

* Patients receiving any other agent or therapy to treat their malignancy
* Pre-existing gastrointestinal disorders which may interfere with absorption of drugs
* Clinically significant cardiovascular disease
* Pregnant or lactating women
* HIV-positive patients receiving combination antiretroviral therapy
* Amendment J and onward for patients in the food effect evaluation and for all subsequent patients if dosing with a high fat/high calorie meal is found to be optimal: Patients with allergies to any ingredient in the defined liquid supplement and/or inability to tolerate a high fat/high calorie meal twice daily on scheduled RO5045337 dosing days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose/Dose-limiting toxicities | approximately 4.5 years
Safety: Incidence of adverse events | approximately 4.5 years
Comparison of daily versus twice daily dosing: Incidence of adverse events | approximately 4.5 years

SECONDARY OUTCOMES:
Pharmacokinetics: Blood/Urine concentrations | Pre- and post-dose multiple sampling Days 1+2/Days 1+10 Cycle 1, post-dose sampling Days 11+15 Cycle 1, pre-dose Days 1+2 Cycle 2
Pharmacodynamics: Blood leukemia cells/MIC-1 protein level/CD33+CD34 markers | Pre- and post-dose Days 1+10 Cycle 1, pre-dose Day 2 Cycle 1, Days 1+2 Cycle 2
Clinical response: Clinical/hematologic malignancy assessments | approximately 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- United States (4):
  - Duarte, California
  - New Brunswick, New Jersey
  - New York, New York
  - Houston, Texas
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- Italy (2):
  - Bologna, Emilia-Romagna
  - Rome, Lazio
- United Kingdom (3):
  - Glasgow
  - Leeds
  - Oxford